CLINICAL TRIAL: NCT02882321
Title: Phase 1 Study of IACS-010759 in Subjects With Relapsed or Refractory AML
Brief Title: Oxidative Phosphorylation Inhibitor IACS-010759 in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor for apparent lack of effectiveness.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0250; NCI-2017-00620 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0250 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — IACS-010759

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 1 (Experimental): IACS-010759 Starting dose: 0.5 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  Interventions: Drug: Oxidative Phosphorylation Inhibitor IACS-010759
- Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 2 (Experimental): IACS-010759 Starting dose: 1 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  Interventions: Drug: Oxidative Phosphorylation Inhibitor IACS-010759
- Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 3 (Experimental): IACS-010759 Starting dose: 2 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of course 1 and on days 1, 8, and 15 of subsequent courses. Treatment repeats every 21 days for subsequent courses for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of oxidative phosphorylation inhibitor IACS-010759 at the discretion of study doctor.
  Interventions: Drug: Oxidative Phosphorylation Inhibitor IACS-010759; Other: Pharmacological Study
- Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 4 (Experimental): IACS-010759 Starting dose: 2.5 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of course 1 and on days 1, 8, and 15 of subsequent courses. Treatment repeats every 21 days for subsequent courses for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of oxidative phosphorylation inhibitor IACS-010759 at the discretion of study doctor.
  Interventions: Drug: Oxidative Phosphorylation Inhibitor IACS-010759; Other: Pharmacological Study

INTERVENTIONS:
Drug: Oxidative Phosphorylation Inhibitor IACS-010759 — Given PO
  Other Names: IACS-010759; OXPHOS Inhibitor IACS-010759
Other: Pharmacological Study — Correlative studies
  Arms: Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 3; Treatment (oxidative phosphorylation inhibitor IACS-010759) Cohort 4

SUMMARY:
This phase I trial studies the side effects and best dose of oxidative phosphorylation inhibitor IACS-010759 in treating patients with acute myeloid leukemia that has come back or does not respond to treatment. Oxidative phosphorylation inhibitor IACS-010759 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined the study. Up to 6 groups of 3-6 participants will be enrolled in the dose escalation part of the study. Up to 18 participants will be enrolled in dose expansion.

OUTLINE: This is a dose-escalation study.

INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 orally (PO) once daily (QD) on days 1-7.

MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of course 1 and on days 1, 8, and 15 of subsequent courses. Treatment repeats every 21 days for subsequent courses for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of oxidative phosphorylation inhibitor IACS-010759 at the discretion of study doctor.

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

If you are enrolled in dose escalation, the dose of IACS-010759 you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of IACS-010759. Each new group will receive a higher dose of IACS-010759 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of IACS-010759 is found.

If you are enrolled in the dose expansion part of the study, you will receive the dose level of IACS-010759 that was found to be the best dose in the escalation part of the study.

In the dose expansion part of the study, 6 participants will also be enrolled in a food-effect group (described in more detail below) to help researchers understand the effects of taking the study drug with food.

Study Drug Administration Each study cycle is 21 days. Cycle 1 only is 28 days. You will take IACS-010759 by mouth one (1) time every day. On Day 1 of Cycle 1 only, you will take your first dose of IACS-010759 and then wait 7 days to take your next dose. Starting on Day 8 of Cycle 1, you will take the study drug every day for the next 21 days.

You will be admitted to the hospital on Day 1 of Cycle 1 for 24 hours and on Day 8 of Cycle 1 for 7 days. This is done so that you can be checked on for any side effects.

Length of Study You may continue to take IACS-010759 for up to 12 cycles. If the doctor thinks it is in your best interest, you may be able to continue receiving the study drug beyond 12 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

ELIGIBILITY:
Inclusion:

1. Subjects with AML should have failed any prior induction therapy regimen or have relapsed after prior therapy (defined as patients in first relapse and less than 12 months from diagnosis [short first remission] or in second or later relapse: Dose-escalation phase: Subjects with confirmed relapsed or refractory AML and no available treatment options with known benefit. Expansion phase: Subjects with relapsed/refractory AML who have failed therapy with up to one prior salvage regimen and no available treatment options with known benefit Exception: SCT or stem cell therapy for subjects who previously underwent SCT/stem cell therapy, and are currently in remission will not be considered a salvage regimen.
2. Eastern Cooperative Oncology Group (ECOG) </= 2
3. Patients who have had prior SCT are eligible if they have a relapse > 3 months since autologous or allogeneic stem cell transplantation provided, 1) No clinically significant active graft-versus-host disease (GVHD > grade 1); 2) No treatment with high dose steroids for GVHD (i.e. >20 mg Prednisolone or equivalent per day); 3) No treatment with immunosuppressive drugs with the exception of cyclosporine and tacrolimus.
4. Subjects with history of central nervous system (CNS) disease are allowed if at the time of day 1 of the study there is no evidence of active CNS disease as documented by negative imaging or spinal fluid analysis carried out at least 2 weeks prior to the first study drug administration in a subject with no clinical signs of CNS disease.
5. Adequate renal and hepatic function: 1) Serum creatinine </= 2.0 X ULN; 2) Total bilirubin </= 2 times the upper limit of normal (ULN) (or </= 3.0 x ULN if deemed to be elevated due to Gilbert's disease or leukemia); 3) Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) </= 2.5 times ULN (</= 5.0 x ULN if due to leukemic involvement).
6. Negative urine pregnancy test within 72 hours prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post- menopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).
7. Have been informed of other treatment options and is not a candidate for standard treatment options or stem cell transplant at the time of enrollment.
8. Age >/= 18 years.
9. In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of IACS-010759 administration will be at least 2 weeks or 5 half-lives (whichever is shorter) for cytotoxic/noncytotoxic agents and biological/immune therapies, including investigational agents. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochures, or drug-administration manuals) and will be documented in the protocol eligibility document. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal therapy for subjects with controlled CNS leukemia at the discretion of the PI and with the agreement of the Sponsor. (2) Use of hydroxyurea for subjects with rapidly proliferative disease is allowed before the start of study therapy and for the first 2 cycles on therapy. These medications will be recorded in the case-report form.
10. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include: 1) Total abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; 2) Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment;
11. #10 continued: 3) Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject;4) Combination of any of the two following (a+b or a+c or b+c): a. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception;b. Placement of an intrauterine device (IUD) or intrauterine system (IUS); c. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository. In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.
12. #11 continued: Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
13. Able and willing to give valid written informed consent.

Exclusion:

1. Prior exposure to IACS-010759 or other oxidative phosphorylation Inhibitors.
2. Unstable cardiovascular function: 1) Symptomatic ischemia, or 2) Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or 3) Congestive heart failure (CHF) NYHA Class >/= 3, or 4) Myocardial infarction (MI) within 6 months; 5) Left ventricular ejection fraction < 40 %; 6) hypertension > 160 mm Hg systolic or > 100 mm Hg diastolic with or without antihypertensive therapy.
3. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery from the surgical procedure
4. Presence of >/= CTCAE grade 2 toxicity (except alopecia or peripheral neuropathy) due to prior cancer therapy.
5. Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV).
6. Active uncontrolled infection. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
7. Participation in any other clinical trial involving another investigational agent for the treatment of AML within 2 weeks prior to day 1 of the study or at least 5 half-lives of the investigational agent, whichever is shorter.
8. Lactate levels > 2 mmol/L and or and serum pH <7.35 at screening.
9. Subject currently being treated with biguanides or other agents known to increase risk of lactic acidosis.
10. Subject has significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhea associated with intestinal malabsorption, Crohn's disease, and/or prior surgical procedures affecting absorption or requirement for intravenous (IV) alimentation.
11. Subjects with uncontrolled Type I or II diabetes mellitus
12. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
13. Women who are breast-feeding or pregnant as evidenced by positive urine pregnancy test done within 72 hours of first dosing.
14. Subject has a concurrent active malignancy under treatment, with the exception of: -Adequately treated carcinoma in situ of the breast or cervix uteri; -Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; -Low-grade, early-stage prostate cancer with no requirement for therapy; -Previous malignancy confined
15. Acute promyelocytic leukemia.
16. Any concomitant disease or condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.
17. Subjects with >/= grade 1 peripheral neuropathy at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yap TA, Daver N, Mahendra M, Zhang J, Kamiya-Matsuoka C, Meric-Bernstam F, Kantarjian HM, Ravandi F, Collins ME, Francesco MED, Dumbrava EE, Fu S, Gao S, Gay JP, Gera S, Han J, Hong DS, Jabbour EJ, Ju Z, Karp DD, Lodi A, Molina JR, Baran N, Naing A, Ohanian M, Pant S, Pemmaraju N, Bose P, Piha-Paul SA, Rodon J, Salguero C, Sasaki K, Singh AK, Subbiah V, Tsimberidou AM, Xu QA, Yilmaz M, Zhang Q, Li Y, Bristow CA, Bhattacharjee MB, Tiziani S, Heffernan TP, Vellano CP, Jones P, Heijnen CJ, Kavelaars A, Marszalek JR, Konopleva M. Complex I inhibitor of oxidative phosphorylation in advanced solid tumors and acute myeloid leukemia: phase I trials. Nat Med. 2023 Jan;29(1):115-126. doi: 10.1038/s41591-022-02103-8. Epub 2023 Jan 19. PMID 36658425
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1: IACS-010759 Starting dose: 0.5 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  Oxidative Phosphorylation Inhibitor IACS-010759: Given PO
- Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2: IACS-010759 Starting dose: 1 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  Oxidative Phosphorylation Inhibitor IACS-010759: Given PO
- Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3: IACS-010759 Starting dose: 2 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of course 1 and on days 1, 8, and 15 of subsequent courses. Treatment repeats every 21 days for subsequent courses for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of oxidative phosphorylation inhibitor IACS-010759 at the discretion of study doctor.
  Oxidative Phosphorylation Inhibitor IACS-010759: Given PO
  Pharmacological Study: Correlative studies
- Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4: IACS-010759 Starting dose: 2.5 mg
  INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of course 1 and on days 1, 8, and 15 of subsequent courses. Treatment repeats every 21 days for subsequent courses for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of oxidative phosphorylation inhibitor IACS-010759 at the discretion of study doctor.
  Oxidative Phosphorylation Inhibitor IACS-010759: Given PO
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
Started | 4 | 3 | 3 | 7
Completed | 4 | 3 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5 | 10
  >=65 years | 2 | 1 | 2 | 2 | 7
Age, Continuous [Median (Full Range); unit: years] | 64 [45 to 71] | 56 [49 to 76] | 70 [60 to 77] | 52 [29 to 77] | 60 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 4 | 7
  Male | 3 | 1 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 5 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Defined as the Highest Dose Studied for Which the Observed Incidence of Dose Limiting Toxicities (DLT) is Less Than 33%
Description: Will be assessed according to National Cancer Institute Common Toxicity Criteria version 4.03.
Time Frame: Up to 28 days
Measure: Number; unit: Milligrams (MG)
Groups:
- Phase I (Cohorts 1-4): INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7.
  Oxidative Phosphorylation Inhibitor IACS-010759: Given PO
Arm/Group | Phase I (Cohorts 1-4)
Number analyzed (Participants) | 17
Milligrams (MG) | NA — The study was terminated before determination of Maximum Tolerated Dose (MTD) was determined.

2. Secondary Outcome: Participants With a Response
Description: Response is Complete Response (CR) + Complete Response with Incomplete Blood Count Recovery (CRi) + Partial Response (PR) + Morphologic Leukemia -Free State (MLFS): CR is Bone marrow blasts < 5%; absence of circulating blasts and blasts with Auer rods; absence of extra-medullary disease; ANC > 1.0 x 10^9/L; platelet count >/= 100 x 10^9/L. CRi is CR except for ANC </= 1.0 x 10^9 or platelet count , 100 x 10^9/L. PR is decreased bone marrow blast % by at least 50% to a value of 5% to 25% and ANC >/= 1.0 x 10^9/L; platelet count >/= 100 x 10^9/L. MLFS is Bone marrow blasts < 5%; abcence of blasts with Auer rods; absence of extra-medullary disease; no hematologic recovery required.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
Number analyzed (Participants) | 4 | 3 | 3 | 7
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of Response
Description: Duration of Response: length of time from the first objective evidence of response to the first objective evidence of disease progression.
Time Frame: Up to 5 years
Population: Zero participants in cohorts 1-4 had a response.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
Number analyzed (Participants) | 4 | 3 | 3 | 7
Months | NA [NA to NA] — Duration of Response can't be calculated as zero participants had a response. | NA [NA to NA] — Duration of Response can't be calculated as zero participants had a response. | NA [NA to NA] — Duration of Response can't be calculated as zero participants had a response. | NA [NA to NA] — Duration of Response can't be calculated as zero participants had a response.

4. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival: length of time (up to 5 years) from the date of first treatment to the first objective evidence of disease progression or death, whichever is earlier.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
Number analyzed (Participants) | 4 | 3 | 3 | 7
Months | 1.3 [0.9 to 1.8] | 1.5 [1.5 to 1.7] | 1.4 [1.1 to 2.8] | 0.5 [0.3 to 1.2]

5. Secondary Outcome: Overall Survival
Description: Overall Survival: length of time from the date of first administration of study drug to the date of death from any cause.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
Number analyzed (Participants) | 4 | 3 | 3 | 7
Months | NA [NA to NA] — Median and full range could not be reached due to insufficient number of participants with events. | 5.6 [2.2 to 8.4] | 2.2 [1.9 to 9.2] | 1.6 [0.4 to 2.6]

ADVERSE EVENTS:
Time Frame: Up to 5 years, 6 months
Arm/Group | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/3 | 1/3 | 3/7
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 3/3 | 4/7
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 (N=4) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 (N=3) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 (N=3) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4 (N=7)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage/Bleeding-Other (Specify) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 2 (3) | 1 (1) | 2 (2) | 3 (4)
Neurology (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syndromes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 1 (N=4) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 2 (N=3) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 3 (N=3) | Treatment (Oxidative Phosphorylation Inhibitor IACS-010759) Cohort 4 (N=7)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypoalbumineia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constitutional Symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
xerostomia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fistula, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Magnesium (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory-Othe (Metabolism and nutrition disorders) | 4 (6) | 3 (3) | 2 (2) | 7 (9)
Muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Neurology-Other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ocular/Visual-Other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain-Other (General disorders) | 2 (8) | 0 (0) | 0 (0) | 2 (5)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syndromes-Other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02882321/Prot_SAP_000.pdf